CLINICAL TRIAL: NCT01460368
Title: A Placebo- and Positive-Controlled Study of the Electrophysiological Effects of a Supratherapeutic Dose of LY2409021 in Healthy Subjects
Brief Title: A Study on the Effects of LY2409021 on the Electrical Impulses of the Heart
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 14149; I1R-FW-GLBP (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-10-07; First posted 2011-10-26 (Estimated); Results first posted 2018-10-18 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — adomeglivant; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part A: LY2409021 (Experimental): Participants will receive 2 standard meals; one alone without LY2409021, and one along with a single dose of 300 milligrams (mg) LY2409021 administered orally. Participants enrolled in Part A will not be allowed to participate in Part B.
  Interventions: Drug: LY2409021
- Part B: LY2409021 (Experimental): 300 milligrams (mg) LY2409021 administered orally as a single dose on Day 1 of the relevant treatment period. The treatment and washout period was a total of 15 days in length.
  Interventions: Drug: LY2409021
- Part B: Placebo (Placebo Comparator): Administered orally as a single dose on Day 1 of the relevant treatment period. The treatment and washout period was a total of 15 days in length.
  Interventions: Drug: Placebo
- Part B: Moxifloxacin (Active Comparator): 400 milligrams (mg) Moxifloxacin administered orally as a single dose on Day 1 of the relevant treatment period. The treatment and washout period was a total of 15 days in length.
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: LY2409021 — Administered orally
  Arms: Part A: LY2409021; Part B: LY2409021
Drug: Placebo — Administered orally
  Arms: Part B: Placebo
Drug: Moxifloxacin — Administered orally
  Arms: Part B: Moxifloxacin

SUMMARY:
Part A: The purpose of Part A of the study is to look at the electrocardiogram (ECG) effects due to blood sugar changes after a meal compared to when LY2409021 is also given with a meal.

Part B: The purpose of Part B is to evaluate the effect of LY2409021, when given at a dose level much higher than what would normally be given, on the electrical activity of the heart as measured by ECG in relation to placebo and moxifloxacin.

DETAILED DESCRIPTION:
This is a 2 part study. Part A is a single-dose study to compare the effects of a meal on glucose, insulin and QT in healthy participants with and without LY2409021. Part B of this study is a randomized, 3-period, crossover design, in which participants and investigators are blinded to placebo and LY2409021, and will assess the electrophysiological effects of a single supratherapeutic dose of LY2409021 compared to a positive control (moxifloxacin) and placebo.

ELIGIBILITY:
Inclusion Criteria:

* are overtly healthy males or females, as determined by medical history and physical examination
* female participants: women not of child-bearing potential due to surgical sterilization (hysterectomy alone or at least 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy or tubal ligation) confirmed by medical history, or menopause Women with an intact uterus are deemed postmenopausal if they are >=45 years old, have not taken hormones or oral contraceptives within the last year, had cessation of menses for at least 1 year, or have had 6 to 12 months of amenorrhea with follicle-stimulating hormone levels consistent with postmenopausal state
* have a body mass index (BMI) of 18.5 to 32 kilograms per meter squared (kg/m^2), inclusive, at screening
* have a fasting blood glucose between 54 to 110 milligrams per deciliter (mg/dL) (3.0 to 6.1 millimoles per liter [mmol/L])
* have a clinically normal screening electrocardiogram (ECG) with a measurable QT interval as judged by central reader, which allows accurate measurements of QT interval
* have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* have venous access sufficient to allow for blood sampling
* are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* have normal blood pressure and pulse rate (supine) at screening, or with minor deviations judged to be acceptable by the investigator
* have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site
* serum magnesium and potassium equal to or above the lower limit of normal

Exclusion Criteria:

* are currently enrolled in or have completed or discontinued within the last 30 days (from screening) from a clinical trial involving an investigational product; or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* have known allergies to LY2409021, related compounds or any components of the formulations, or to moxifloxacin
* are persons who have previously received the investigational product in this study, have completed or withdrawn from this study or any other study investigating LY2409021
* personal or family history of long QT syndrome
* family history of sudden unexplained death or cardiac death in a family member under 60 years of age
* personal history of unexplained syncope within the last year
* have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* show evidence of hepatitis C and/or positive hepatitis C antibody
* show evidence of hepatitis B and/or positive hepatitis B surface antigen
* are women with a positive pregnancy test or women who are lactating
* intend to use over-the-counter (including mineral supplements and herbal medicine) or prescription medication within 7 days prior to dosing
* have donated blood of more than 500 milliliters (mL) within the last month
* have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females) (1 unit = 12 ounces [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits), or are unwilling to comply with alcohol restrictions during the study (that is, refrain from alcohol consumption from 24 hours prior to dosing until the completion of each treatment period and to consume no more than 2 units of alcohol per day between treatment periods)
* are participants who smoke more than 10 cigarettes per day and/or are unable to abide by the study restrictions for smoking/tobacco use (that is, refrain from smoking for approximately 2 hours prior to each ECG timepoint or for a total of approximately 12 hours)
* are participants who are unable to abide by the study restrictions for caffeine/xanthine use (that is, refrain from consuming caffeine/xanthine containing drinks and foods [such as coffee, tea, cola, and chocolate] on days on which ECGs are performed, and maintain consistent consumption habits on all other days of the study)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: LY2409021: Participants received 2 standard meals; one alone without LY2409021, and one along with a single dose of 300 milligrams (mg) LY2409021 administered orally to determine the effects of a meal on electrocardiogram (ECG) activity. Participants enrolled in Part A were not allowed to participate in Part B.
- Part B: LY2409021, Placebo, Moxifloxacin: Period 1: 300 milligrams (mg) LY2409021 administered orally as a single dose on Day 1.
  Period 2: Placebo administered orally as a single dose on Day 1.
  Period 3: 400 milligrams (mg) Moxifloxacin administered orally as a single dose on Day 1.
- Part B: Moxifloxacin, LY2409021, Placebo: Period 1: 400 milligrams (mg) Moxifloxacin administered orally as a single dose on Day 1.
  Period 2: 300 milligrams (mg) LY2409021 administered orally as a single dose on Day 1.
  Period 3: Placebo administered orally as a single dose on Day 1.
- Part B: Placebo, Moxifloxacin, LY2409021: Period 1: Placebo administered orally as a single dose on Day 1.
  Period 2: 400 milligrams (mg) Moxifloxacin administered orally as a single dose on Day 1.
  Period 3: 300 milligrams (mg) LY2409021 administered orally as a single dose on Day 1.
- Part B: Moxifloxacin, Placebo, LY2409021: Period 1: 400 milligrams (mg) Moxifloxacin administered orally as a single dose on Day 1.
  Period 2: Placebo administered orally as a single dose on Day 1.
  Period 3: 300 milligrams (mg) LY2409021 administered orally as a single dose on Day 1.
- Part B: Placebo, LY2409021, Moxifloxacin: Period 1: Placebo administered orally as a single dose on Day 1.
  Period 2: 300 milligrams (mg) LY2409021 administered orally as a single dose on Day 1.
  Period 3: 400 milligrams (mg) Moxifloxacin administered orally as a single dose on Day 1.
- Part B: LY2409021, Moxifloxacin, Placebo: Period 1: 300 milligrams (mg) LY2409021 administered orally as a single dose on Day 1.
  Period 2: 400 milligrams (mg) Moxifloxacin administered orally as a single dose on Day 1.
  Period 3: Placebo administered orally as a single dose on Day 1.
Period: Part A
Arm/Group | Part A: LY2409021 | Part B: LY2409021, Placebo, Moxifloxacin | Part B: Moxifloxacin, LY2409021, Placebo | Part B: Placebo, Moxifloxacin, LY2409021 | Part B: Moxifloxacin, Placebo, LY2409021 | Part B: Placebo, LY2409021, Moxifloxacin | Part B: LY2409021, Moxifloxacin, Placebo
Started | 7 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 7 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B: First Intervention (Period 1)
Arm/Group | Part A: LY2409021 | Part B: LY2409021, Placebo, Moxifloxacin | Part B: Moxifloxacin, LY2409021, Placebo | Part B: Placebo, Moxifloxacin, LY2409021 | Part B: Moxifloxacin, Placebo, LY2409021 | Part B: Placebo, LY2409021, Moxifloxacin | Part B: LY2409021, Moxifloxacin, Placebo
Started | 0 | 10 | 10 | 10 | 10 | 10 | 10
Received at Least One Dose of Study Drug | 0 | 10 | 10 | 10 | 10 | 10 | 10
Completed | 0 | 10 | 10 | 10 | 9 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Part B: Washout (up to 15 Days)
Arm/Group | Part A: LY2409021 | Part B: LY2409021, Placebo, Moxifloxacin | Part B: Moxifloxacin, LY2409021, Placebo | Part B: Placebo, Moxifloxacin, LY2409021 | Part B: Moxifloxacin, Placebo, LY2409021 | Part B: Placebo, LY2409021, Moxifloxacin | Part B: LY2409021, Moxifloxacin, Placebo
Started | 0 | 10 | 10 | 10 | 9 | 10 | 10
Completed | 0 | 10 | 10 | 10 | 9 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B: Second Intervention (Period 2)
Arm/Group | Part A: LY2409021 | Part B: LY2409021, Placebo, Moxifloxacin | Part B: Moxifloxacin, LY2409021, Placebo | Part B: Placebo, Moxifloxacin, LY2409021 | Part B: Moxifloxacin, Placebo, LY2409021 | Part B: Placebo, LY2409021, Moxifloxacin | Part B: LY2409021, Moxifloxacin, Placebo
Started | 0 | 10 | 10 | 10 | 9 | 10 | 10
Completed | 0 | 8 | 10 | 10 | 9 | 10 | 9
Not Completed | 0 | 2 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Part B: Washout (up to 15 Days)
Arm/Group | Part A: LY2409021 | Part B: LY2409021, Placebo, Moxifloxacin | Part B: Moxifloxacin, LY2409021, Placebo | Part B: Placebo, Moxifloxacin, LY2409021 | Part B: Moxifloxacin, Placebo, LY2409021 | Part B: Placebo, LY2409021, Moxifloxacin | Part B: LY2409021, Moxifloxacin, Placebo
Started | 0 | 8 | 10 | 10 | 9 | 10 | 9
Completed | 0 | 8 | 9 | 10 | 9 | 10 | 9
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Part B: Third Interventions (Period 3)
Arm/Group | Part A: LY2409021 | Part B: LY2409021, Placebo, Moxifloxacin | Part B: Moxifloxacin, LY2409021, Placebo | Part B: Placebo, Moxifloxacin, LY2409021 | Part B: Moxifloxacin, Placebo, LY2409021 | Part B: Placebo, LY2409021, Moxifloxacin | Part B: LY2409021, Moxifloxacin, Placebo
Started | 0 | 8 | 9 | 10 | 9 | 10 | 9
Completed | 0 | 8 | 8 | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug (Part A or Part B).
Groups:
- Part A: A single dose of 300 milligrams (mg) LY2409021 administered orally on Day 1. Participants enrolled in Part A were not allowed to participate in Part B.
- Part B: Participants received a single dose of either 300 milligrams (mg) LY2409021, 400 mg Moxifloxacin, or Placebo on Day 1 in 1 of 3 Study Periods so that after the completion of the 3 study periods, each participant received a single dose of each drug.
- Total: Total of all reporting groups
Arm/Group | Part A | Part B | Total
Number analyzed (Participants) | 7 | 60 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (7.7) | 39.7 (12.8) | 40.4 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 14 | 14
  Male | 7 | 46 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 20 | 23
  Not Hispanic or Latino | 4 | 40 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 23 | 26
  White | 4 | 35 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 60 | 67

OUTCOME MEASURES:

1. Primary Outcome: Part B: Mean Change From Baseline in 12-lead Electrocardiogram (ECG) Corrected QT Intervals (LY2409021)
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave and was calculated from electrocardiogram (ECG) data using Fridericia's formula: QTc = QT/RR^0.33. Corrected QT (QTc) is the QT interval corrected for heart rate and RR, which is the interval between two R waves. Least Squares (LS) means were calculated using mixed effects model with fixed effects for treatment, time, period, sequence, and the time-by-treatment interaction, random effects for participant, the participant-by-treatment interaction, and participant-by-time interaction.
Time Frame: Baseline, 2, 4, 6, 8, 12, and 24 hours
Population: Participants who received at least 1 dose of LY2409021 or Placebo with evaluable Fridericia Correction Formula (QTcF) data.
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Groups:
- Part B: LY2409021: 300 milligrams (mg) LY2409021 administered orally as a single dose on Day 1 of the relevant treatment period.
- Part B: Placebo: Placebo: Administered orally as a single dose on Day 1 of the relevant treatment period.
Arm/Group | Part B: LY2409021 | Part B: Placebo
Number analyzed (Participants) | 58 | 56
milliseconds
  2 hours postdose: number analyzed (Participants) | 57 | 54
  2 hours postdose | -14.72 [-16.44 to -13.00] | -15.35 [-17.10 to -13.59]
  4 hours postdose: number analyzed (Participants) | 57 | 53
  4 hours postdose | -5.43 [-7.15 to -3.72] | -9.12 [-10.89 to -7.35]
  6 hours postdose: number analyzed (Participants) | 56 | 54
  6 hours postdose | 6.13 [4.40 to 7.85] | -3.01 [-4.77 to -1.26]
  8 hours postdose | 7.80 [6.09 to 9.51] | -1.29 [-3.02 to 0.45]
  12 hours postdose: number analyzed (Participants) | 58 | 55
  12 hours postdose | -13.45 [-15.15 to -11.74] | -13.30 [-15.05 to -11.55]
  24 hours postdose: number analyzed (Participants) | 57 | 55
  24 hours postdose | -1.32 [-3.04 to 0.40] | -4.95 [-6.70 to -3.20]
Statistical Analysis 1: Comparison: Part B: LY2409021 vs Part B: Placebo; Test type: Superiority or Other; Least Squares Mean Difference = 0.63, 90% CI 2-sided [-1.38 to 2.63] — Treatment comparison at 2 hours
Statistical Analysis 2: Comparison: Part B: LY2409021 vs Part B: Placebo; Test type: Superiority or Other; Least Squares Means Difference = 3.69, 90% CI 2-sided [1.67 to 5.71] — Treatment comparison at 4 hours
Statistical Analysis 3: Comparison: Part B: LY2409021 vs Part B: Placebo; Test type: Superiority or Other; Least Squares Means Difference = 9.14, 90% CI 2-sided [7.12 to 11.16] — Treatment comparison at 6 hours
Statistical Analysis 4: Comparison: Part B: LY2409021 vs Part B: Placebo; Test type: Superiority or Other; Least Squares Means Difference = 9.08, 90% CI 2-sided [7.10 to 11.07] — Treatment comparison at 8 hours
Statistical Analysis 5: Comparison: Part B: LY2409021 vs Part B: Placebo; Test type: Superiority or Other; Least Squares Means Difference = -0.15, 90% CI 2-sided [-2.14 to 1.85] — Treatment comparison at 12 hours
Statistical Analysis 6: Comparison: Part B: LY2409021 vs Part B: Placebo; Test type: Superiority or Other; Least Squares Means Difference = 3.63, 90% CI 2-sided [1.63 to 5.63] — Treatment comparison at 24 hours

2. Secondary Outcome: Part B: Mean Change From Baseline in 12-lead Electrocardiogram (ECG) Corrected QT Intervals (Moxifloxacin)
Description: as for outcome 1
Time Frame: Baseline, 2 and 4 hours
Population: Participants who received at least 1 dose of Moxifloxacin or Placebo with evaluable QTcF data.
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Groups:
- Part B: Moxifloxacin: 400 milligrams (mg) Moxifloxacin administered orally as a single dose on Day 1 of the relevant treatment period.
Arm/Group | Part B: Moxifloxacin | Part B: Placebo
Number analyzed (Participants) | 56 | 54
milliseconds
  2 hours postdose: number analyzed (Participants) | 55 | 54
  2 hours postdose | -7.39 [-9.13 to -5.64] | -15.46 [-17.22 to -13.70]
  4 hours postdose: number analyzed (Participants) | 56 | 53
  4 hours postdose | 1.45 [-0.28 to 3.18] | -9.11 [-10.88 to -7.34]
Statistical Analysis 1: Comparison: Part B: Moxifloxacin vs Part B: Placebo; Test type: Superiority or Other; Least Squares Mean Difference = 8.07, 90% CI 2-sided [5.21 to 10.94] — Treatment comparison at 2 hours
Statistical Analysis 2: Comparison: Part B: Moxifloxacin vs Part B: Placebo; Test type: Superiority or Other; Least Squares Mean Difference = 10.56, 90% CI 2-sided [7.69 to 13.43] — Treatment comparison at 4 hours

ADVERSE EVENTS:
Groups:
- Part A: LY2409021: A single dose of 300 milligrams (mg) LY2409021 administered orally on Day 1. Participants enrolled in Part A were not allowed to participate in Part B.
- Part B: Placebo: Administered orally as a single dose on Day 1 of the relevant treatment period.
Arm/Group | Part A: LY2409021 | Part B: Placebo | Part B: Moxifloxacin | Part B: LY2409021
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/57 | 0/58 | 0/59
Other Adverse Events (participants affected / at risk) | 1/7 | 12/57 | 11/58 | 9/59
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: LY2409021 (N=7) | Part B: Placebo (N=57) | Part B: Moxifloxacin (N=58) | Part B: LY2409021 (N=59)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Application site rash (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Application site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hangnail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days